CLINICAL TRIAL: NCT03165383
Title: The Analgesic Efficacy of Ultrasound Guided Transversus Abdominis Plane (TAP) Block in Lower Abdominal OncoSurgeries
Brief Title: The Analgesic Efficacy of Ultrasound Guided Transversus Abdominal Plane Block After Abdominal Cancer Surgeries
Acronym: TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr Anita Kulkarni, Principal Investigator, Rajiv Gandhi Cancer Institute & Research Center, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGCI & RC
Record Dates: First submitted 2017-05-18; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Abdominal Cancer
Keywords: Transverse Abdominis Plane (TAP) Block; Patient Control Analgesia (PCA)
MeSH Terms: conditions — Bites and Stings | interventions — Bupivacaine; Analgesia, Patient-Controlled; Passive Cutaneous Anaphylaxis; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversus Abdominis Plane (TAP) Block Group (Active Comparator): Intervention - At the end of surgery Ultrasound guided Transversus Abdominis Plane block was given with 20 ml 0.25 % bupivacaine bolus and repeated every 8 hourly upto 24 hours.
  Interventions: Drug: Bupivacaine (Transversus Abdominis Plane Block)
- Control Group (No TAP Block) (Placebo Comparator): The Transversus Abdominis Plane Block was not performed. Intravenous PCA Morphine was given as rescue analgesic upto 24 hours.
  Interventions: Drug: Intravenous Patient Controlled Analgesia (PCA) Morphine

INTERVENTIONS:
Drug: Bupivacaine (Transversus Abdominis Plane Block) — Intervention - At the end of surgery Ultrasound guided Transversus Abdominis Plane block was given with 20 ml 0.25 % bupivacaine bolus and repeated every 8 hourly up to 24 hours.
  Arms: Transversus Abdominis Plane (TAP) Block Group
Drug: Intravenous Patient Controlled Analgesia (PCA) Morphine — PCA Intravenous Morphine 1 milligram bolus on demand was given as rescue analgesia up to 24 hours.
  Arms: Control Group (No TAP Block)

SUMMARY:
Effective postoperative pain control results in decreased cardiac and pulmonary complications, patient satisfaction and early mobilization. A prospective, randomized comparative study was done of analgesic efficacy, opioid requirement and side effects in patients undergoing lower abdominal cancer surgeries. In Study Group Ultrasound guided Transversus Abdominis Plane (TAP) block was given and control Group no TAP block was given. Patient controlled analgesia (PCA) with intravenous morphine was given to both group patients, and total good PCA demands in both the groups was studied.

DETAILED DESCRIPTION:
Adult patients of both sexes undergoing major lower abdominal cancer surgeries were enrolled in the study. After obtaining written informed consent from all the patients, they were randomly allotted to either Study (TAP) Group or Control group. Standard general anesthesia with endotracheal intubation was performed in all the patients. Preoperatively all patients received information about Visual Analogue Scale (VAS) for Pain Score from 1 to 10 depending on intensity of pain and about the use of Patient Controlled Analgesia (PCA) Pump. After the end of surgery and before extubation bilateral Ultrasound guided Transversus Abdominis Plane (TAP) block was performed with 16 G Tuohy needle and 18 G Braun Perifix epidural catheter was placed about 6-8 cms in situ. Bupivacaine 0.25 % 20 ml was given bilaterally and repeated 8 hourly in the Postoperative Anaesthesia Care Unit (PACU) for first 24 hours. The PCA Pump was set to deliver bolus Intravenous Morphine 1 milligram ( mg ) with lock out interval 10 minutes. In the PACU heart rate, Non invasive blood pressure, Visual Analogue Score at rest and on knee flexion, Sedation score, nausea and vomiting, any side effects as itching was noted by care provider at 0, 2, 4, 6, 12, 18 and 24 hours. Total and good PCA demands upto 24 hours was recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients belonging to American Society of Anesthesiologist (ASA) Physical Status I to III, for Open lower abdominal major onco surgeries more than 2 hours duration.

Exclusion Criteria:

* Patient refusal to participate in the study, allergy to local anesthetics, coagulopathy, local skin infection at the site of TAP Block.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02-11 (Actual); Primary Completion 2014-07-10 (Actual); Study Completion 2014-08-20 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Pain Score in PACU in Transversus Abdominis Plane Block and Control Patient Group. | up to 24 hours
  In the PACU Visual Analogue Pain Score will be noted at rest and on knee flexion up to 24 hours.

SECONDARY OUTCOMES:
Total and Good demands for PCA IV Morphine in milligrams in both the groups. | up to 24 hours
  In the PACU, Total and Good PCA IV Morphine demands in milligrams in both groups was studied.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kulkarni, MD, Principal Investigator — Rajiv Gandhi Cancer Institute and Research Centre , Delhi , India 110085

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158
- [Result] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269